CLINICAL TRIAL: NCT06311110
Title: Impaired Toilet Training, Lower Urinary Tract Symptoms and Bowel Dysfunction in Children With Developmental Coordination Disorder
Brief Title: Impaired Toilet Training, LUTS and Bowel Dysfunction in Children With DCD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: #BC-11326 AM04
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Developmental Coordination Disorder; Lower Urinary Tract Symptoms; Bowel Dysfunction
MeSH Terms: conditions — Motor Skills Disorders; Lower Urinary Tract Symptoms; Intestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DCD case group: The case group consists of children with developmental coordination disorder.
  Interventions: Other: Vancouver symptom score for dysfunctional elimination symptoms Questionnaire; Other: Developmental Coordination Disorder Questionnaire; Other: Questionnaire concerning impaired toilettraining and comorbities
- TDC control group: The control group consists of typically developing children, grade and gender matched with the DCD case group.
  Interventions: Other: Vancouver symptom score for dysfunctional elimination symptoms Questionnaire; Other: Developmental Coordination Disorder Questionnaire; Other: Questionnaire concerning impaired toilettraining and comorbities

INTERVENTIONS:
Other: Vancouver symptom score for dysfunctional elimination symptoms Questionnaire — Vancouver symptom score for dysfunctional elimination syndrome, Dutch version, validated by 't Hoen et al. 2016. The questionnaire is filled in by the parents of the child.
  Other Names: VSSDES
Other: Developmental Coordination Disorder Questionnaire — Validated Developmental Coordination Disorder Questionnaire, Dutch version includes assessment of motor functioning. The questionnaire is filled in by the parents of the child.
  Other Names: DCD-Q; CVO
Other: Questionnaire concerning impaired toilettraining and comorbities — Unvalidated, complementary questions concerning impaired toilettraining and comorbidities. Questions were based on ICCS standardisation guidelines (Austin et al., 2015). The questionnaire is filled in by the parents of the child.

SUMMARY:
This cross-sectional case-control study aimed to determine whether there is a significant difference in the prevalence of impaired toilet training, LUTS, and functional bowel problems among children diagnosed with DCD and typically developing children (TDC).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DCD by a multidisciplinary team (DCD case group)
* Children with a typical development, grade and gender matched with the DCD case group (TDC control group).

Exclusion Criteria:

* A DCD-Q score indicative for DCD (TDC control group)
* Presence of other developmental disorders, such as ASS, ADHD or intellectual disability (TDC control group)

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with developmental coordination disorder and grade- and gender matched typically developing children.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Impaired toilet training | through study completion, 25 minutes
  Prevalence of impaired toilet training in children with DCD compared to TDC
Daytime incontinence | through study completion, 25 minutes
  Prevalence of daytime incontinence at 5 years old in children with DCD compared to TDC
Enuresis | through study completion, 25 minutes
  Prevalence of enuresis at 5 years old in children with DCD compared to TDC
Fecal incontinence | through study completion, 25 minutes
  Prevalence of fecal incontinence at 4 years old in children with DCD compared to TDC

SECONDARY OUTCOMES:
Toilet training difficulties | through study completion, 25 minutes
  Prevalence and amount of toilet training difficulties in children with DCD compared to TDC
General bladder and bowel dysfunction | through study completion, 25 minutes
  Prevalence of LUTS, bowel problems or combined bladder and bowel dysfunction in children with DCD compared to TDC

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Vandamme, MD, Principal Investigator — University Hospital, Ghent; Bieke Samijn, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital/Ghent University, Ghent, East Flanders
  - University Hospital Ghent, Ghent